CLINICAL TRIAL: NCT06860984
Title: Evaluating the Safety and Efficacy of Duloxetine in the Prevention of Post Endoscopic Retrograde Cholangiopancreatography Pancreatitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5487
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Biliary Disease
MeSH Terms: conditions — Gallbladder Diseases | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): The patients will receive placebo capsule placebo tablet 2 h before ERCP.
  Interventions: Other: Placebo capsule
- Duloxetine group (Active Comparator): The patients will receive 60 mg duloxetine 2 h before ERCP.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Duloxetine, a non-opioid neuromodulator, has been widely used to manage neuropathic pain. It possesses dual central and peripheral analgesic properties
  Arms: Duloxetine group
Other: Placebo capsule — Placebo will have the same look and appearance of active comparator
  Arms: Control group

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP (, a key tool that is used in diagnosis and treatment of pancreato-biliary diseases. Post-ERCP pancreatitis (PEP) is the most common and serious complication that can occur following this procedure and can lead to significant morbidity and mortality. A variety of patient-related and procedure-related factors have been associated with higher rates of PEP.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old.
* Gender: Males and Females
* Patients with suitable indications for ERCP due to suspected pancreato-biliary disorders.
* Blood amylase and lipase levels before ERCP are within the normal limits

Exclusion Criteria:

* Uncontrolled diabetes mellitus (DM)
* Severe bleeding tendency
* Impaired renal function (serum creatinine > 2 mg/dL), (creatinine clearance <30 ml/min)
* Patients with severe heart disease.
* Subjects who underwent prior biliary or pancreatic sphincterotomy or dilatation or stenting of either duct.
* Currently pregnant or nursing
* Admission due to established pancreatitis before ECRP
* Unwillingness to undergo ERCP.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
The primary outcome that will be measured is the development of pancreatitis after the procedure | 24 hours
  The primary outcome that will be measured is the development of pancreatitis after the procedure according to consensus criteria. Briefly in this criteria PEP will be diagnosed if the Patient met two of the three following criteria after ERCP: new onset or increased abdominal pain consistent with acute pancreatitis, pancreatic enzyme elevation to at least 3 times the upper limit of normal at 24 hours after the procedure, and the necessity for new or continued hospitalization for at least 2 nights.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt